CLINICAL TRIAL: NCT06499675
Title: Prevalence of Steatosis and Steatohepatitis in Patients Undergoing Bariatric Surgery; a Biopsy-based Study
Status: Completed | Type: Observational
Sponsor: Egyptian Liver Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Steatosis2019
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Obesity, Morbid; Bariatric Surgery Candidate; Steatosis of Liver; Steatohepatitis, Nonalcoholic
Keywords: steatosis; bariatric surgery; liver biopsy
MeSH Terms: conditions — Obesity; Obesity, Morbid; Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver Biopsy slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: obese patients
  Interventions: Procedure: sleeve gastrectomy; Procedure: Liver Biopsy

INTERVENTIONS:
Procedure: sleeve gastrectomy — sleeve gastrectomy / bariatric surgery
Procedure: Liver Biopsy — intraoperative liver biopsy

SUMMARY:
To study the prevalence of steatosis, steatohepatitis, and their associated risk factors in obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
A prospective single-center biopsy-based study was conducted on 162 sleeve gastrectomy patients. Patient characteristics, including age, sex, diabetes mellitus (DM) status, body mass index (BMI), liver function tests, lipogram, homeostatic model assessment of insulin resistance (HOMA-IR), and steatosis were also assessed using controlled attenuation parameter (CAP), and intra operative liver biopsies were obtained. , The presence of steatosis and steatohepatitis were histologically assessed by two expert pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic sleeve gastrectomy ≥18 years of age.
* Able to give written informed consent.
* Scheduled, independently from this study, to have a liver biopsy (LB).
* Negative for hepatitis B surface antigen, anti-hepatitis C virus, hepatitis C virus-RNA, and hepatitis B virus DNA.
* BMI greater than or equal to 40, or BMI greater than or equal to 35 with at least one obesity-related comorbid condition (including type 2 diabetes, hypertension, hyperlipidemia, obstructive sleep apnea (OSA), GERD, asthma, venous stasis disease, severe osteoarthritis, or considerably impaired quality of life).
* Unsuccessful nonoperative weight loss attempts.
* Mental health clearance.
* Recent updates have included patients with a BMI of 30-35 with uncontrollable type 2 diabetes or metabolic syndrome as an indication for a laparoscopic sleeve gastrectomy.

Exclusion Criteria:

* Patients with ascites.
* Pregnant women.
* Patients with any active implantable medical device (such as pacemaker or defibrillator).
* Patients who had undergone liver transplantation.
* Patients with cardiac failure and significant valvular disease.
* Patients with hemochromatosis.
* Patients who refused to undergo liver biopsy or blood tests.
* Patients with alcohol consumption above recommended limits (>14 units/week for women and >21 units/week for men; 1 unit = 8 g of ethanol).
* Patients with a confirmed diagnosis of active malignancy or another terminal disease.
* Patients participating in another clinical trial within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a cross-sectional prospective single-center study conducted between May 2019 and December 2023.
  The study included consecutive patients receiving sleeve gastrectomy at the Egyptian Liver Research Institute and Hospital (ELRIAH), Sherbin, El-Mansoura, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Compare the histological assessment of steatosis and steatohepatitis with non invasive procedures. | 55 months
  Compare the histological assessment of steatosis and steatohepatitis with non invasive procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Liver Research Institute and Hospital (ELRIAH), Sherbin, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided